CLINICAL TRIAL: NCT03043547
Title: A Randomized Phase II Trial of Nal-IRI and 5-Fluorouracil Compared to 5-Fluorouracil in Patients With Cholangio- and Gallbladder Carcinoma Previously Treated With Gemcitabine-based Therapies
Brief Title: Nal-IRI and 5-FU Compared to 5-FU in Patients With Cholangio- and Gallbladder Carcinoma Previously Treated With Gemcitabine-based Therapies
Acronym: NALIRICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-HEP-0116; 2016-003709-33 (EudraCT Number)
Record Dates: First submitted 2017-01-26; First posted 2017-02-06 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cholangiocarcinoma Non-resectable; Cholangiocarcinoma Metastatic; Cholangiocarcinoma of the Gallbladder; Cholangiocarcinoma Advanced
Keywords: nal-IRI; 5-Fluorouracil
MeSH Terms: interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nal-IRI + 5-FU + leucovorin (Arm A) (Experimental): nal-IRI [Irinotecan liposome] (80 mg/m2 as a 1.5 hour infusion), 5-FU [5-Fluorouracil] (2400 mg/m2 as 46 hour infusion) and leucovorin (400 mg/m2 as 0.5 hour infusion) (q2w)
  Interventions: Drug: nal-IRI; Drug: 5-FU; Drug: leucovorin
- 5-FU + leucovorin (Arm B) (Other): Control intervention/standard arm: 5-FU (2400 mg/m2 as 46 hour infusion) and leucovorin (400 mg/m2 as 0.5 hour infusion) (q2w)
  Interventions: Drug: 5-FU; Drug: leucovorin

INTERVENTIONS:
Drug: nal-IRI — nal-IRI [Irinotecan liposome] (80 mg/m2 as a 1.5 hour infusion)
  Arms: Nal-IRI + 5-FU + leucovorin (Arm A)
Drug: 5-FU — 5-FU [5-Fluorouracil] (2400 mg/m2 as 46 hour infusion)
Drug: leucovorin — leucovorin (400 mg/m2 as 0.5 hour infusion)

SUMMARY:
is an open label, randomized, multicenter phase II trial

DETAILED DESCRIPTION:
The primary objective is to assess the efficacy of nal-IRI in gemcitabine pre-treated patients with advanced, unresectable and metastatic cholangio- and gallbladder carcinoma eligible for treatments after failure to respond to a gemcitabine-based treatment

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent incl. participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Histologically or cytologically confirmed, non-resectable, locally advanced or metastatic cholangiocarcinoma or gall bladder carcinoma
4. Measurable or assessable disease according to RECIST 1.1
5. Documented disease progression after prior gemcitabine or gemcitabine containing therapy, in locally advanced or metastatic setting. Examples of permitted therapies include, but are not limited to:

   1. Single agent gemcitabine
   2. Any one gemcitabine-based regimen, with or without maintenance gemcitabine
6. ECOG performance status 0-1
7. Adequate blood count, liver-enzymes, and renal function:

   * ANC > 1,500 cells/μL without the use of hematopoietic growth factors; and
   * Platelet count ≥ 100 x 10^9/L (>100,000 per mm³) and
   * Hemoglobin > 9 g/dL (blood transfusions are permitted for patients with hemoglobin levels below 9 g/dL)
   * Serum total bilirubin ≤ 3x upper normal limit (ULN) (biliary drainage is allowed for biliary obstruction; elevated bilirubin should be caused by obstruction not impaired liver function as assessed by albumin and INR values):
   * Albumin levels ≥ 3.0 g/dL
   * Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and PTT < 1.5 ULN within 7 days prior to randomization. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of randomization
   * AST (SGOT)/ALT (SGPT) ≤ 5 x institutional upper limit of normal
   * Serum Creatinine ≤ 1.5 x ULN and a calculated glomerular filtration rate ≥ 30 mL per minute
8. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of treatment.
9. Subject is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Active CNS metastases (indicated by clinical symptoms, cerebral oedema, steroid requirement, or progressive disease); patient should have been off steroids for at least 28 days prior to starting study therapy
2. Clinically significant gastrointestinal disorder including bleeding, inflammation, occlusion, or diarrhoea > grade 1
3. History of any second malignancy in the last 5 years; subjects with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible. Subjects with other malignancies are eligible if they have been continuously disease free for at least 5 years.
4. Active uncontrolled infection, chronic infectious diseases, immune deficiency syndromes or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, patients with tumour fever may be enrolled), which in the investigator's opinion might compromise the patient's participation in the trial or affect the study outcome.
5. Premalignant hematologic disorders, e.g. myelodysplastic syndrome
6. Pre-existing lung disease
7. Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 6 months before enrollment
8. History of hypersensitivity to any of the study drugs or any excipient (nal-IRI, other liposomal products, fluoropyrimidines or leucovorin)
9. Allogeneic transplantation requiring immunosuppressive therapy or other major immunosuppressive therapy
10. Severe non-healing wounds, ulcers or bone fractions
11. Evidence of bleeding diathesis or coagulopathy
12. Major surgical procedures, except open biopsy, nor significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgical procedure during the course of the study except for surgery of central intravenous line placement for chemotherapy administration.
13. Medication that is known to interfere with any of the agents applied in the trial.
14. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are:implants, injectable contraceptives, combined oral contraceptives, intrauterine pessaries (only hormonal devices), sexual abstinence or vasectomy of the partner].
15. Known Gilbert-Meulengracht syndrome
16. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
17. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 5 half-lifes of previously used trial medication, whichever is of longer duration.
18. Previous enrollment or randomization in the present study (does not include screening failure).
19. Previous enrollment in the NIFE trial [AIO-YMO/HEP-0315]
20. Involvement in the planning and/or conduct of the study (applies to both Baxalta staff and/or staff of sponsor and study site)
21. Patient who might be dependent on the sponsor, site or the investigator
22. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
23. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
progression-free survival | approx 42 months

SECONDARY OUTCOMES:
Overall survival | approx 42 months
Objective tumor response rate (ORR) according to RECIST 1.1 | approx 42 months
  Response Evaluation Criteria in Solid Tumors (RECIST 1.1.)
Toxicity/Safety | approx 42 months
  according to Common Terminology Criteria for Adverse Events
Health related Quality of Life | approx 42 months
  EORTC QLQ-C30

OTHER OUTCOMES:
biomarkers | approx 42 months
  Ca-19-9, CEA, CRP serum levels
Immunohistochemistry of Carboxylesterase (CES) | approx 42 months
Analyse whole blood | approx 42 months
  will be collected to potentially identify factors that may correlate with tumour response, sensitivity or resistance to nal-IRI
Analyse plasma | approx 42 months
  will be collected to potentially identify factors that may correlate with tumour response, sensitivity or resistance to nal-IRI

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Vogel, Prof., Principal Investigator — Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Medizinische Hochschule Hannover
Locations (1):
- Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Medizinische Hochschule Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoo C, Saborowski A, Hyung J, Wenzel P, Kim I, Wege H, Kim KP, Folprecht G, Ryoo BY, Schutt P, Cheon J, Gotze T, Ryu H, Lee JS, Vogel A. Liposomal irinotecan for previously treated patients with biliary tract cancer: A pooled analysis of NIFTY and NALIRICC trials. J Hepatol. 2025 Oct;83(4):909-916. doi: 10.1016/j.jhep.2025.03.013. Epub 2025 Mar 25. PMID 40147791
- [Derived] Vogel A, Saborowski A, Wenzel P, Wege H, Folprecht G, Kretzschmar A, Schutt P, Jacobasch L, Ziegenhagen N, Boeck S, Zhang D, Kanzler S, Belle S, Mohm J, Gokkurt E, Lerchenmuller C, Graeven U, Pink D, Gotze T, Kirstein MM. Nanoliposomal irinotecan and fluorouracil plus leucovorin versus fluorouracil plus leucovorin in patients with cholangiocarcinoma and gallbladder carcinoma previously treated with gemcitabine-based therapies (AIO NALIRICC): a multicentre, open-label, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2024 Aug;9(8):734-744. doi: 10.1016/S2468-1253(24)00119-5. Epub 2024 Jun 10. PMID 38870977
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de/projekte.html